CLINICAL TRIAL: NCT04078607
Title: Effect of a Cognitive Distraction on Amount, Preference, and Memory of Food Consumed: a Randomized Crossover Exploratory Study
Brief Title: Cognitive Distraction on Food Intake: Randomized Crossover Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Shelly Nickols-Richardson, Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: liguori
Record Dates: First submitted 2019-08-18; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Obesity; Weight, Body
Keywords: Distraction; Eating behavior; Fullness; Hunger; Ingestive behavior; Rapid visual information processing
MeSH Terms: conditions — Obesity; Body Weight; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled crossover study where participants were assigned to begin in the distracted or control condition. One week later, participants completed the opposite condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distraction (Experimental): Distraction during eating using the Rapid Visual Information Processing task as the distraction
  Interventions: Behavioral: Rapid Visual Information Processing task
- Control (Placebo Comparator): No distraction during eating
  Interventions: Behavioral: None or Control condition

INTERVENTIONS:
Behavioral: Rapid Visual Information Processing task — A series of numbers appeared on a computer screen at a rate of one per minute. Each participant was required to identify any series of three consecutive odd or even numbers by hitting the space bar on the keyboard. The task lasted 15 minutes and included a 1-minute practice session before food being served. Participants were instructed to eat at will while completing the computer task.
  Arms: Distraction
Behavioral: None or Control condition — Participant were instructed to eat at will during a 15-minute duration.
  Arms: Control

SUMMARY:
This study determined effects of a cognitive distraction on amount, preference, and memory of food consumed and perceptions of fullness, hunger, and enjoyment of food in a healthy young-adult population. A randomized controlled crossover study of 119 healthy adults, assigned to begin in either the distracted or control condition, was conducted.

DETAILED DESCRIPTION:
Environmental distractions have been shown to affect eating patterns. Influences of food environments on consumption patterns and not simply food choices are becoming increasingly clear for their contributions to energy intake. Of particular interest is the presence of distraction. It has been postulated that when distracted, individuals are inclined to consumer more than when not distracted. However, how distraction and memory impact subsequent food choice and preference is less well known. A Rapid Visual Information Processing (RVIP) task was applied to distract individuals while eating; food intake and food behaviors were measured after RVIP distraction and compared to food intake and food behaviors without distraction in the same individuals.

ELIGIBILITY:
Inclusion Criteria:

* able to read and speak English and willing to consume foods provided during the study

Exclusion Criteria:

* adhering to any dietary restrictions or diets, having any food allergies, and/or having any chronic or metabolic diseases

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Food intake | Up to 14 days
  Consumption of food by number of food items eaten

SECONDARY OUTCOMES:
Snack intake | Up to 14 days
  Consumption of snack choices by number of food items eaten
Memory of food intake | Up to 14 days
  Recording of food that was eaten during the condition period by number of food items eaten
Fullness | Up to 14 days
  How full do you feel right now? by 100mm visual analog scale; 0=not at all to 100=very much
Hunger | Up to 14 days
  How hungry do you feel right now? by 100mm visual analog scale; 0=not at all to 100=very much
Enjoyment | Up to 14 days
  How much did you enjoy the meal provided? by 100mm visual analog scale; 0=not at all to 100=very much

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Nickols-Richardson, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared if required by journal requirements and/or as requested by other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately until after publication of study
Access Criteria: Contact with the primary investigator using criteria of co-publishing, collaborating on same topic, or using data as preliminary findings for further studies; primary investigator will review requests

REFERENCES:
- [Derived] Liguori CA, Nikolaus CJ, Nickols-Richardson SM. Cognitive Distraction at Mealtime Decreases Amount Consumed in Healthy Young Adults: A Randomized Crossover Exploratory Study. J Nutr. 2020 May 1;150(5):1324-1329. doi: 10.1093/jn/nxaa022. PMID 32060552